CLINICAL TRIAL: NCT05381597
Title: Combination of 5-Fluorouracil and Calcipotriene in the Treatment of Superficial Basal Cell Carcinomas and Squamous Cell Carcinomas in Situ
Brief Title: 5-Fluorouracil and Calcipotriene for Treatment of Low Grade Skin Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-42421
Record Dates: First submitted 2022-05-15; First posted 2022-05-19 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Superficial Basal Cell Carcinoma; Squamous Cell Carcinoma in Situ
Keywords: 5-fluorouracil cream; fluorouracil with calcipotriene
MeSH Terms: conditions — Squamous Intraepithelial Lesions | interventions — calcipotriene

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Combination cream of 5-fluorouracil and calcipotriene (Experimental): Participants randomized to this group will receive treatment with the combination cream consisting of 5-fluorouracil and calcipotriene twice a day for 7 days and the treatment can be extended to 14 days based on evaluation at 7 days.
  Interventions: Drug: Combination cream of 5-fluorouracil and calcipotriene
- 5-fluorouracil cream (Active Comparator): Participants randomized to this group will receive treatment with 5-fluorouracil cream twice a day for 28 days.
  Interventions: Drug: 5-fluorouracil cream

INTERVENTIONS:
Drug: Combination cream of 5-fluorouracil and calcipotriene — Apply the cream to the size of the lesion extending to the 0.5 cm area of skin surrounding the lesion.twice a day for 7 days and the treatment can be extended to 14 days based on evaluation at 7 days.
  Other Names: compounded cream
  Arms: Combination cream of 5-fluorouracil and calcipotriene
Drug: 5-fluorouracil cream — Apply the cream to the size of their lesion extending to the 0.5 cm area of skin surrounding the lesion twice daily for 28 days.
  Other Names: usual treatment
  Arms: 5-fluorouracil cream

SUMMARY:
The investigators will compare the application of two different creams for the treatment of low-risk skin cancers-superficial basal cell carcinoma (sBCC) and squamous cell carcinoma in situ (SCCis). 5-Fluorouracil cream is currently FDA approved for the treatment of superficial basal cell carcinoma and is routinely used by dermatologists across the country and at Boston Medical Center (BMC) for SCCis. The normal treatment regimen is 4 weeks of the 5-fluorouracil cream for both skin cancers.

The application of a compounded cream consisting of 1:1 ratio 5-fluorouracil with calcipotriene will be tested. This combination cream has been shown to clear pre-skin cancers called actinic keratoses and prevent future skin cancers from developing. This combination cream for 7-14 days to see if this shorter treatment course provides clearance of the 2 types of skin cancer. This combination cream is successfully used in this manner to treat other subtypes of related skin cancers. This will be a pilot study with

The primary endpoint for this pilot randomized single blinded clinical trial will be the response to treatment (yes versus no). The lesions will be assessed clinically for clearance of cancer, as would normally be done and is consistent with how comparable studies have assessed clearance. Participants will be followed closely afterwards for three years with visits at 6 months, which does not vary from standard practice. If the lesions are not clear of cancer or equivocal clinically, the lesions will be re-biopsied and normal standard of care procedure will take place.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Having a previously untreated, biopsy-proven Superficial Basal Cell Carcinoma (sBCC) or Squamous Cell Carcinoma in Situ (SCCis) of the skin <2 cm on the scalp, trunk, neck, or extremities, excluding hands, feet, and genitalia
* Having a previously untreated, biopsy-proven sBCC or SCCis on the face, hands, feet, and genitalia who decline surgery or are otherwise not surgical candidates
* Willing to undergo all protocol requirements and attend study-specific follow up clinic visits in addition to routine follow up visits
* Participants may have multiple lesions enrolled in the study so long as the individual lesions are greater than 2 cm from each other
* If a woman is of childbearing potential, the participant must be willing to take a pregnancy test before starting treatment and be on some form of birth control while receiving treatment. Birth control can include abstinence, oral contraceptive pill, intrauterine device, implanted birth control device, birth control patch, or the vaginal ring. The patient does not need to be on any form of birth control after they end therapy.

Exclusion Criteria:

* Current or prior field treatment within 2 cm of the target BCC or SCCis
* Periorbital lesions
* Lesions that have been previously treated
* Known allergy to any of the study medication ingredients
* History of solid organ transplant or current immunosuppression
* Genetic disorders associated with high skin cancer risk
* Arsenic exposure
* Cutaneous T-cell lymphoma
* Current or prior radiation therapy at the site of the sBCC or SCCis
* Women who are pregnant or currently breastfeeding
* Prior psoralen plus Ultraviolet light (UVA) treatment at the site
* Very high mortality risk at the start of the study
* Dihydropyrimidine dehydrogenase (DPD) enzyme deficiency
* Demonstrated hypercalcemia or evidence of vitamin D toxicity
* Lesions that extend into the oral, nasal or genital mucosa

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Clearance rate of cancer lesions at 3 months | 3 months
  Clearance rate is defined as the percentage of lesions that are free of cancer based on clinical assessments which will be performed by the patient's dermatologist and via photos from a standardized full frontal angle.
Clearance rate of cancer lesions at 3 years | 3 years
  Clearance rate is defined as the percentage of lesions that are free of cancer based on clinical assessments which will be performed by the patient's dermatologist and via photos from a standardized full frontal angle.

SECONDARY OUTCOMES:
Percent of participants that experience pain during treatment | 3 months
  Based on responses to an investigator-developed survey completed by each participant within 5 days of treatment completion, participants will rate their pain from 1 to 5 where 1=no pain, 2= very mild, 3=mild, 4=moderate (requiring pain medication), 5=severe (requiring pain medication or physician contact). The number of participants with scores of 2 or higher will be divided by all participants.
Severity of pain during treatment | 3 months
  Based on responses to an investigator-developed survey completed by each participant within 5 days of treatment completion, participants will rate their pain from 1 to 5 where 1=no pain, 2= very mild, 3=mild, 4=moderate (requiring pain medication), 5=severe (requiring pain medication or physician contact). Mean pain ratings will be calculated with higher mean scores suggesting more severe pain.
Percent of participants that experience redness during treatment | 3 months
  Based on responses to an investigator-developed survey completed by each participant within 5 days of treatment completion, participants will rate their overall redness from 1 to 5 where 1=no redness, 2= very minimal, 3=minimal, 4=moderate, 5=severe. The number of participants with scores of 2 or higher will be divided by all participants.
Severity of redness during treatment | 3 months
  Based on responses to an investigator-developed survey completed by each participant within 5 days of treatment completion, participants will rate their overall redness from 1 to 5 where 1=no redness, 2= very minimal, 3=minimal, 4=moderate, 5=severe. Mean redness ratings will be calculated with higher mean scores suggesting more severe redness.
Day of worst redness | 3 months
  For participants who experienced any redness, the mean day after treatment when the redness was worst will be calculated.
Percent of participants who experienced scaling/flaking | 3 months
  Based on responses to an investigator-developed survey completed by each participant within 5 days of treatment completion, participants will be asked if they experienced any scaling/flaking. The number of participants who responded 'yes' will be divided by all participants.
Percent of participants who experienced skin itching | 3 months
  Based on responses to an investigator-developed survey completed by each participant within 5 days of treatment completion, participants will be asked if they experienced any skin itching. The number of participants who responded 'yes' will be divided by all participants.
Percent of participants who experienced skin burning | 3 months
  Based on responses to an investigator-developed survey completed by each participant within 5 days of treatment completion, participants will be asked if they experienced any skin burning. The number of participants who responded 'yes' will be divided by all participants.
Participant compliance with treatment | 3 months
  Compliance with treatment will be assessed by weighing the medicine tubes after treatment completion and comparing the weight, estimated in grams from fingertip units (FTU), with the expected weight based on the how much medicine should have been used given the treatment regimen. The closer this difference is to zero, the greater the compliance.
Participant satisfaction with treatment | 3 months
  Based on responses to an investigator-developed survey completed by each participant within 5 days of treatment completion, participants will rate their satisfaction with the treatment from 1 to 5 where 1=very dissatisfied, 2= dissatisfied, 3=neutral, 4=satisfied, 5=very satisfied. Mean satisfaction ratings will be calculated with higher mean scores suggesting more treatment satisfaction.
Recurrence rate of cancer lesions at 1 year | 1 year
  The recurrence rate is the percentage of cancer lesions that recur which is the number that recur out of the number cleared.
Recurrence rate of cancer lesions at 3 years | 3 years
  The recurrence rate is the percentage of cancer lesions that recur which is the number that recur out of the number cleared.

CONTACTS AND LOCATIONS:
Overall Officials: Bilal Fawaz, MD, Principal Investigator — Dermatology, Boston University School of Medicine
Locations (1):
- Boston Medical Center Dermatology Clinic, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No